CLINICAL TRIAL: NCT00481923
Title: A Randomized, Double-Bind, Placebo-Controlled, Parallel-Group, Fixed-Dose (20 mg/Day), 3-Month, Multicenter Study of the Energy Intake Effects and Safety of SR141716 With or Without Hypocaloric Diet in Obese Patients
Brief Title: Efficacy and Safety of Rimonabant With or Without Hypocaloric Diet in Obese Patients
Acronym: REBA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5031
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Obesity
Keywords: hypocaloric diet; energy intake
MeSH Terms: conditions — Obesity | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rimonabant (SR141716)

SUMMARY:
The primary objective of this study is to assess the effect of rimonabant on the energy intake (kcal/day/meal) from ad-libitum high-fat dinner (primary endpoint), pre- and post-ingestive responses, and the hedonic evaluation of food, and its effect on food choice, cravings and feelings of control.

The secondary objectives are to determine the effect of rimonabant on body weight with or without hypocaloric diet and its clinical and laboratory safety.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects with Body Mass Index ≥ 30 and < 45 kg/m²

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2004-05; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in energy intake during ad-libitum dinner of the high-fat probe day at Weeks 3/4 of double-blind treatment.

SECONDARY OUTCOMES:
Satiety, food choice, feeling of control, craving using a series of rating scales during the probe and/or "free-living" days
Clinical Safety

CONTACTS AND LOCATIONS:
Overall Officials: John Blundell, Pr, Principal Investigator — University of Leeds, United Kingdom
Locations (1):
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom